CLINICAL TRIAL: NCT04597996
Title: The Effect of Web-Based Mental Health Literacy Program on Students' Level of Knowledge, Help-Seeking and Stigmatization Attitudes
Brief Title: Web-based Mental Health Literacy Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, ozlem ozkan salkim, Public Health Nursing PhD student, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/23-23
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Mental Health Literacy
Keywords: Web Based; Health Education; School Nurse; Mental Health Literacy; Adolescents; Students
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: pre test post test model design
Who Masked: Participant
Masking Description: students
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web Based Education (Experimental): A pre-test will be applied. Web-based education will be conducted. The post-test will be applied twice, the first one to be performed 4 weeks after Web-based education is completed and the second one 3 months after Web-based education is completed.
  Interventions: Other: web based education for students
- No Intervention Group (No Intervention): The control group will not have any intervention during the study.

INTERVENTIONS:
Other: web based education for students — Web-based education will include modules on the following subjects;
  * Mental health literacy knowledge level
  * Improving help-seeking behavior
  * Avoiding self-stigmatization in seeking psychological help
  Arms: Web Based Education

SUMMARY:
Mental health literacy is a concept that aims to improve the skills of individuals to overcome difficulties in providing the appropriate help they need in this area. It provides individuals with motivation in this area such as informing and taking responsibility in the field of mental health, directing their behavior, facilitating access to and obtaining information, understanding, evaluating, using, and maintaining information.

Objective: This project aims to examine the effect of web-based mental health literacy intervention carried out by school nurses on students' level of knowledge, help-seeking and stigmatization attitudes.

Method: Randomized Controlled Trial Research design (pre-test post-test control group design) will be used in the project. The data will be collected through the Mental Health Literacy Scale for Children and Adolescents (MHLS), Attitude Scale for Seeking Psychological Help-Short Form (ASPH-S), Self-Stigma in Seeking Psychological Help Scale (SSSPHS) and the sociodemographic Question Form.

The project will be carried out with the students of a secondary school and a high school in the district of Balçova, İzmir province. Sampling calculation Based on the analysis of variance in repeated measurements in 2 groups in the G Power program, Type1 Error 0.05 (alpha 5%) Type2 Error 0.20 (80% power), the sample size calculated in duplicate measurements with medium effect size is 43 participants for each group (Intervention-Control) calculated. Considering that there might be losses during data collection, it is planned to include 50 students for the intervention group and 50 students for the control group. Analysis of variance will be used in the evaluation of data, number, percentage, and descriptive statistics, and in repeated measures to evaluate the effect of the intervention The training modules to be prepared within the scope of the project will focus on the mental health literacy level of the child, attitudes to seek help and stigmatization. Among the teaching materials planned to be prepared for this purpose, there will be short animated course videos, video course contents, and audio presentations. In the study, where web-based education is planned, teaching materials will be delivered to students through the learning management system. Teaching materials and learning management systems will be designed in accordance with mobile technologies and access will be provided from smartphones, tablet computers, and similar mobile devices. During the teaching material development phase, firstly, educational content drafts (storyboards) will be created and presented to field experts, and their opinions on content, teaching approach, methods and techniques, and visual design principles will be taken. Pilot studies will be conducted to understand the educational content during the improvement phase of the developed teaching material designs. It is planned to finalize the training content in light of user feedback.

DETAILED DESCRIPTION:
In this study, the investigators aim to examine the effect of mental health literacy Web-based education intervention on the knowledge level, help-seeking and stigmatization attitudes of students.

This study is a randomized controlled trial. The study population consists of students studying in two schools located in Izmir province in western Turkey. Fifty people were assigned to the intervention and control groups each and a total of 100 participants were planned to be included.

The study will be conducted between January-September 2022. Students between the ages of 12-18 who voluntarily agree to participate in the study will be included in this study. Another criterion is that all sampled groups be able to access and use the internet.

Those who have visual, perceptual, or auditory problems and cannot access or use the internet will not be included in the study.

Psychometric evaluation of scales:

Mental Health Literacy Scale for Children and Adolescents (MHLS): This scale, developed by Rozbruch and Friedberg (2018), consists of 5 items. The Cronbach alpha coefficient calculated for the internal consistency of the scale is .84. The scale is a three-point Likert-type scale consisting of two items multiple choice, one item open-ended, two items 8 sub-dimensions (Parents, Friends, Clergyman, Psychologist, Counselor, Psychiatrist, Family Doctor, Teacher) (not suitable - not sure - suitable) has the option to answer. The lowest value that can be taken from the scale varies between 0 and the highest value: 6. (question 1: 1 point, question 3: 2 points, question 4: 2 points, question 5: 1 point) Turkish adaptation of the scale was made by the researchers Attitude Scale for Seeking Psychological Help-Short Form (ASPH-S): This tool, which aims to measure attitudes towards getting psychological help (ASPH-S), is a revised and abbreviated version of ASPH, developed by Türküm (1997). As a result of the factor analysis performed for the construct validity of the ASPH-S scale, it was determined that it consists of a two-factor structure that includes positive (12 items) and negative (6 items) seeking psychological help, explaining 52.6% of the total variance. The Cronbach's alpha coefficient calculated for internal consistency of the scale consisting of 18 items is .90. Test-retest reliability for stability over time. It was found to be 77. The score that can be obtained from the scale is between 18 and 90, and the low score indicates that there is no need for help. The scale, which consists of 5 Likert-type categories, is scored as Fully Agree, Strongly Agree, Undecided, Somewhat Agree, and Never Disagree. (Fully Agree = 5, Strongly Agree = 4, Undecided = 3 Somewhat Agree = 2, Not at all = 1) 6 items of the scale are calculated by scoring in reverse. These items are: 2, 8, 12, 13, 16, 17.

Self-Stigma in Seeking Psychological Help Scale (SSSPHS): The scale developed by Vogel et al. (2006) consists of ten items. The scale is a 5-point Likert type one-dimensional scale. The scale was adapted to Turkish by Kapıkıranlar (2013). Cronbach alpha value is calculated for the internal consistency of the scale. Is 71. Confirmatory factor analysis of the one-dimensional scale was performed. The internal consistency of university students (17-33) was calculated as .91, and the test-retest reliability with an interval of two months was calculated as .72. Some items of the scale are scored reversely, and high scores indicate the high level of self-stigma in asking for help. Some items of the scale are scored inversely, and a high score indicates a high level of self-stigma in asking for help.

Ethics Committee approval was obtained from Dokuz Eylül University Health Sciences Institute. (2019 / 23-23) The permit of the institution will be obtained from the İzmir Provincial Directorate of the National Education Strategy Development Unit. Informed consent will be obtained from the parents on behalf of their children.

Dependent Variable: Adolescent Mental Health Literacy knowledge level, Attitudes towards Seeking Psychological Help, Self-Stigma in Seeking Psychological Help score averages

Independent Variable: Mental Health literacy education

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 12-18 (inclusive)
* volunteering to participate
* having the access to internet
* knowing how to use the internet
* without visual impairment
* without hearing impairment
* without perceptual impairment

Exclusion Criteria:

* not volunteering to participate
* not having the access to internet
* not knowing how to use the internet
* with visual impairment
* with hearing impairment
* with perceptual impairment

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Mental Health Literacy Scale for Children and Adolescents (MHLS) | 3 MONTH
  It is a three-point Likert-type scale consisting of two items multiple choice, one item open-ended, two items 8 sub-dimensions (Parents, Friends, Clergyman, Psychologist, Counselor, Psychiatrist, Family Doctor, Teacher) (not suitable - not sure - suitable) has the option to answer. The lowest value that can be taken from the scale varies between 0 and the highest value: 6. (question 1: 1 point, question 3: 2 points, question 4: 2 points, question 5: 1 point).
Attitude Scale for Seeking Psychological Help-Short Form (ASPH-S) | 3 MONTH
  It consists of a two-factor structure that includes positive (12 items) and negative (6 items) seeking psychological help, explaining 52.6% of the total variance. The scale, which consists of 5 Likert-type categories, is scored as Fully Agree, Strongly Agree, Undecided, Somewhat Agree, and Never Disagree. (Fully Agree = 5, Strongly Agree = 4, Undecided = 3 Somewhat Agree = 2, Not at all = 1) 6 items of the scale are calculated by scoring in reverse. These items are: 2, 8, 12, 13, 16, 17.The score that can be obtained from the scale is between 18 and 90, and the low score indicates that there is no need for help.
Self-Stigma in Seeking Psychological Help Scale (SSSPHS) | 3 MONTH
  The scale is a 5-point Likert type one-dimensional scale with 10 items. Some items of the scale are scored reversely, and high scores indicate the high level of self-stigma in asking for help. Some items of the scale are scored inversely, and a high score indicates a high level of self-stigma in asking for help.

CONTACTS AND LOCATIONS:
Overall Officials: ozlem ozkan salkim, Principal Investigator — Dokuz Eylul University; Seyda OZBICAKCI, Assoc. Prof, Study Director — Dokuz Eylul University; Yasemin KAHYAOĞLU ERDOĞMUŞ, PhD, Principal Investigator — Dokuz Eylul University

IPD SHARING:
Plan to Share IPD: No